CLINICAL TRIAL: NCT00342732
Title: The Food Intake Phenotype: Assessing Eating Behavior and Food Preferences as Risk Factors for Obesity
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999019; OH99-DK-N019
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-15

CONDITIONS: Obesity; Overweight; Overnutrition
Keywords: Genetics; Fat Intake; Weight Control; Appetite Control; Natural History
MeSH Terms: conditions — Obesity; Overweight; Overnutrition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-diabetic volunteers: non-diabetic volunteers aged 18-65 who are healthy as determined by medical history, physical examination, and laboratory tests

SUMMARY:
The prevalence of obesity in the United States has reached alarming proportions with 33% of adults over the age of 20 being overweight. Obesity is more than twice as prevalent, however, in the Pima Indians of Arizona. Although there have been a number of advances in our understanding of the genetics of obesity, the environmental influences on the genetic expression of obesity requires further investigation.

In an effort to understand some of the influences on the high prevalence of obesity in the Pima Indians, the present study was designed to investigate eating behaviors and food preferences, most especially the preference for high fat foods, in sib-pairs of Pima Indians who have been previously genotyped in our genomic scan for loci linked to diabetes/obesity. Most specifically, we will utilize several questionnaires and methods of assessing eating behavior and the preference for high fat foods to create a food intake phenotype. In addition, we will study Caucasians so that comparisons can be made between these two groups. We will make these evaluations by assessing eating behavior, food preferences including usual fat intake and preferences for high fat foods, body image perceptions, and energy expenditure. It is hoped that the data gathered from this study will elucidate some of the risk factors for the development of obesity among the Pima Indians....

DETAILED DESCRIPTION:
The prevalence of obesity in the United States has reached alarming proportions with 33% of adults over the age of 20 being overweight. In some populations, obesity is even more prevalent. Although there have been a number of advances in our understanding of the genetics of obesity, the environmental influences on the genetic expression of obesity requires further investigation.

In an effort to understand some of the influences on the high prevalence of obesity, the present study was designed to investigate what drives how much people eat. More specifically, we will try to understand what drives food intake utilizing 1) questionnaires that assess eating behavior, 2) measurements in blood, urine or fat tissue, and 3) genotypic associations to investigate the various factors that control what and how much people eat. We will make these evaluations by assessing eating behavior, food preferences including usual fat intake and preferences for high fat foods, body image perceptions, and energy expenditure. It is hoped that the data gathered from this study will elucidate some of the risk factors for the development of obesity.

ELIGIBILITY:
* Inclusion Criteria:

  1. Healthy, as determined by medical history, physical examination, and laboratory tests.
  2. 18-65 years old
  3. Non-diabetic status

Exclusion Criteria:

1. Hypo- or hyper-thyroid
2. Blood pressure greater than 160/95
3. Cardiovascular disease
4. Gallbladder disease
5. Alcohol and/or current use of drugs (more than 2 drinks per day and regular use of drugs such as amphetamines, cocaine, or heroin)
6. Psychiatric conditions or behavior that would be incompatible with safe and successful participation in this study, including claustrophobia and eating disorders such as anorexia or bulimia nervosa

8. Use of medications affecting metabolism and appetite

9. Pregnancy

10. Current use of nicotine products, including tobacco, electronic cigarettes, and nicotine replacement therapies that exceed Very Low Dependence on the Fagerstr(SqrRoot)(Delta)m Test for Nicotine Dependence Tool (score greater than 2).

Subjects may be excluded or withdrawn from the study if they have any conditions not specifically mentioned above that may interfere with the collection of the food intake. This includes such issues as not following study and unit policies and procedures, diagnosis of contraindications following admission, and development of illness/infection unrelated to the study. For example, volunteers who do not comply with the vending machine protocol (i.e., share food, do not record what they eat, eat outside of room, etc) may be withdrawn from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Phoenix metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 669 (Actual)
Dates: Start 1999-11-24 (Actual)

PRIMARY OUTCOMES:
Ad libitum food intake | Baseline, up to day 3
  Ad libitum food intake measured in kcal/day averaged over 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Votruba, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aydin BN, Stinson EJ, Cabeza De Baca T, Ando T, Travis KT, Piaggi P, Krakoff J, Chang DC. Investigation of seasonality of human spontaneous physical activity and energy expenditure in respiratory chamber in Phoenix, Arizona. Eur J Clin Nutr. 2024 Jan;78(1):27-33. doi: 10.1038/s41430-023-01347-y. Epub 2023 Oct 13. PMID 37833567
- [Derived] Booker JM, Chang DC, Stinson EJ, Mitchell CM, Votruba SB, Krakoff J, Gluck ME, Cabeza de Baca T. Food insecurity is associated with higher respiratory quotient and lower glucagon-like peptide 1. Obesity (Silver Spring). 2022 Jun;30(6):1248-1256. doi: 10.1002/oby.23437. PMID 35674698
- [Derived] Cabeza de Baca T, Piaggi P, Gluck ME, Krakoff J, Votruba SB. Meal-to-meal and day-to-day macronutrient variation in an ad libitum vending food paradigm. Appetite. 2022 Apr 1;171:105944. doi: 10.1016/j.appet.2022.105944. Epub 2022 Jan 21. PMID 35074459
- [Derived] Basolo A, Hollstein T, Shah MH, Walter M, Krakoff J, Votruba SB, Piaggi P. Higher fasting plasma FGF21 concentration is associated with lower ad libitum soda consumption in humans. Am J Clin Nutr. 2021 Oct 4;114(4):1518-1522. doi: 10.1093/ajcn/nqab204. PMID 34159373
- [Derived] Basolo A, Ando T, Chang DC, Hollstein T, Krakoff J, Piaggi P, Votruba S. Reduced Albumin Concentration Predicts Weight Gain and Higher Ad Libitum Energy Intake in Humans. Front Endocrinol (Lausanne). 2021 Mar 11;12:642568. doi: 10.3389/fendo.2021.642568. eCollection 2021. PMID 33776937
- [Derived] Hollstein T, Basolo A, Ando T, Votruba SB, Krakoff J, Piaggi P. Urinary Norepinephrine Is a Metabolic Determinant of 24-Hour Energy Expenditure and Sleeping Metabolic Rate in Adult Humans. J Clin Endocrinol Metab. 2020 Apr 1;105(4):1145-56. doi: 10.1210/clinem/dgaa047. PMID 32002540
- [Derived] Stinson EJ, Graham AL, Thearle MS, Gluck ME, Krakoff J, Piaggi P. Cognitive dietary restraint, disinhibition, and hunger are associated with 24-h energy expenditure. Int J Obes (Lond). 2019 Jul;43(7):1456-1465. doi: 10.1038/s41366-018-0305-9. Epub 2019 Jan 16. PMID 30651576
- [Derived] Stinson EJ, Votruba SB, Venti C, Perez M, Krakoff J, Gluck ME. Food Insecurity is Associated with Maladaptive Eating Behaviors and Objectively Measured Overeating. Obesity (Silver Spring). 2018 Dec;26(12):1841-1848. doi: 10.1002/oby.22305. Epub 2018 Nov 14. PMID 30426695
- [Derived] Basolo A, Heinitz S, Stinson EJ, Begaye B, Hohenadel M, Piaggi P, Krakoff J, Votruba SB. Fasting glucagon-like peptide 1 concentration is associated with lower carbohydrate intake and increases with overeating. J Endocrinol Invest. 2019 May;42(5):557-566. doi: 10.1007/s40618-018-0954-5. Epub 2018 Oct 3. PMID 30284224
- [Derived] Stinson EJ, Piaggi P, Ibrahim M, Venti C, Krakoff J, Votruba SB. High Fat and Sugar Consumption During Ad Libitum Intake Predicts Weight Gain. Obesity (Silver Spring). 2018 Apr;26(4):689-695. doi: 10.1002/oby.22124. Epub 2018 Mar 4. PMID 29504262
- [Derived] Stinson EJ, Krakoff J, Gluck ME. Depressive symptoms and poorer performance on the Stroop Task are associated with weight gain. Physiol Behav. 2018 Mar 15;186:25-30. doi: 10.1016/j.physbeh.2018.01.005. Epub 2018 Jan 9. PMID 29326031
- [Derived] Basolo A, Votruba SB, Heinitz S, Krakoff J, Piaggi P. Deviations in energy sensing predict long-term weight change in overweight Native Americans. Metabolism. 2018 May;82:65-71. doi: 10.1016/j.metabol.2017.12.013. Epub 2018 Jan 3. PMID 29305947
- [Derived] Ibrahim M, Thearle MS, Krakoff J, Gluck ME. Perceived stress and anhedonia predict short-and long-term weight change, respectively, in healthy adults. Eat Behav. 2016 Apr;21:214-9. doi: 10.1016/j.eatbeh.2016.03.009. Epub 2016 Mar 3. PMID 27002703
- [Derived] Piaggi P, Thearle MS, Krakoff J, Votruba SB. Higher Daily Energy Expenditure and Respiratory Quotient, Rather Than Fat-Free Mass, Independently Determine Greater ad Libitum Overeating. J Clin Endocrinol Metab. 2015 Aug;100(8):3011-20. doi: 10.1210/jc.2015-2164. Epub 2015 Jun 18. PMID 26086330
- [Derived] Bundrick SC, Thearle MS, Venti CA, Krakoff J, Votruba SB. Soda consumption during ad libitum food intake predicts weight change. J Acad Nutr Diet. 2014 Mar;114(3):444-449. doi: 10.1016/j.jand.2013.09.016. Epub 2013 Dec 8. PMID 24321742
- [Derived] He J, Votruba S, Pomeroy J, Bonfiglio S, Krakoff J. Measurement of ad libitum food intake, physical activity, and sedentary time in response to overfeeding. PLoS One. 2012;7(5):e36225. doi: 10.1371/journal.pone.0036225. Epub 2012 May 22. PMID 22629311
- [Derived] Venti CA, Votruba SB, Franks PW, Krakoff J, Salbe AD. Reproducibility of ad libitum energy intake with the use of a computerized vending machine system. Am J Clin Nutr. 2010 Feb;91(2):343-8. doi: 10.3945/ajcn.2009.28315. Epub 2009 Nov 18. PMID 19923376
- [Derived] Votruba SB, Kirchner H, Tschop M, Salbe AD, Krakoff J. Morning ghrelin concentrations are not affected by short-term overfeeding and do not predict ad libitum food intake in humans. Am J Clin Nutr. 2009 Mar;89(3):801-6. doi: 10.3945/ajcn.2008.27011. Epub 2009 Jan 21. PMID 19158212